CLINICAL TRIAL: NCT02858752
Title: Memory, Auditory and Visual Attention in Healthy Children: Neurophysiological and Electrophysiological Aspects
Brief Title: Memory and Attention in Healthy Children
Acronym: MASK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0711
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
Keywords: Attention; Short-term memory; Aural Memory; Visual Memory; Child; EEG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Children (Experimental): Memory and Attention in healthy children will be assessed non-invasively through behavioral and electrophysiological measures while participants will perform passive or active computer task involving auditory and/or visual perception.
  Interventions: Other: Experience 1 : Auditory and Visual Discrimination; Other: Experience 2 : Passive and Active Auditory Perception; Other: Experience 3 : Visual Attention Training; Other: Experience 4 : Attention and Distractibility; Other: Experience 5 : Sustained Visual Attention

INTERVENTIONS:
Other: Experience 1 : Auditory and Visual Discrimination — Neuropsychological tests consist in listening to sounds in various contexts and providing behavioral responses with response-buttons.
Other: Experience 2 : Passive and Active Auditory Perception — Neuropsychological tests consist in listening to sounds under 2 conditions, an active or a passive one, during which different auditory stimuli will be presented: frequent stimuli (standard) and rare stimuli (deviants). These two stimuli differ in some of their feature (height, duration, …). A third, very rare (novel) stimulus will also be used (the subject's first name). Responses will be provided using a response-button and feedback will be given at each response. EEG will be recorded all along to measure Neurophysiological signals.
Other: Experience 3 : Visual Attention Training — This experience aims at training visual attention through serious games. Children will play against an artificial intelligence and will focus their attention on one out of many possible targets (checkers, cards, boxes) presented on screen. Responses will be provided using a response-button, sometimes completed by an eye-tracking measure. Feedback will be given to the child after his response. EEG will be recorded all along to measure Neurophysiological signals.
Other: Experience 4 : Attention and Distractibility — Neuropsychological tests consist in listening to sounds preceded by a visual cue indicating (or not) in which ear the sounds will be played. The subject Child should detect the target sound (e.g. a dog barking). In some trials, a distracting distraction will be introduced between the visual cue and the target sound. Responses will be provided using a response-button. EEG will be recorded all along to measure Neurophysiological signals.
Other: Experience 5 : Sustained Visual Attention — Neuropsychological tests consist in watching visual stimuli presented in 3 blocks of 3 minutes each, with a break of one minute between each block. The child has to detect the presence of a red letter in a pattern made of four letters (the three other letters are black). Behavioral responses will be provided using a response-button. EEG will be recorded all along to measure Neurophysiological signals.

SUMMARY:
This project studies memory and attention in healthy children aged from 5 to 17 years. The processes investigated are short term memory (auditory and visual) and attention.

To characterize these processes involved in childhood, neuropsychological and neurophysiological assessments will be performed (using Electro-encephalography measures, behavioural responses and questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected vision
* No neurological and psychiatric antecedent.
* No neuro-developmental disorder (dysphasia, dyslexia, dyspraxia, attention deficit disorder…)
* Motivation to participate to the study
* Signed parental informed consent authorizing their child to participate to the study

Exclusion Criteria:

* Children educated in a specialized institution.
* Subjects diagnosed with a neurological, psychiatric or neuro-developmental disorder
* Subjects with hearing loss
* Subjects with a visual impairment that cannot be corrected
* Subjects with an organic or chronic disease that can affect cognitive functions.
* Subjects who do not benefit from social security.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2016-10-06 (Actual); Primary Completion 2020-10-06 (Estimated); Study Completion 2020-10-06 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological tests: Proportion of accurate answers | 2 months
Neuropsychological tests: reaction time of answers (seconds) | 2 months
Neurophysiological tests: Event-related potentials in response to auditory and visual stimulations | 2 months

SECONDARY OUTCOMES:
Proportion of accurate answers according to age range of children | 2 months
reaction time of answers (seconds) according to age range of children | 2 months
Event-related potentials in response to auditory and visual stimulations according to age range of children | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Lyon, France

IPD SHARING:
Plan to Share IPD: No